CLINICAL TRIAL: NCT00921024
Title: A Multicenter, Double-blind, Randomized, Phase 2 Study to Compare the Safety and Efficacy of Intravenous CXA-101 and Intravenous Ceftazidime in Complicated Urinary Tract Infection, Including Pyelonephritis
Brief Title: Safety and Efficacy of IV CXA-101 and IV Ceftazidime in Patients With Complicated Urinary Tract Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7625-001; CXA 101-03 (Other: Cubist Study Number)
Record Dates: First submitted 2009-06-12; First posted 2009-06-16 (Estimated); Results first posted 2015-01-15 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-09

CONDITIONS: Complicated Urinary Tract Infection
Keywords: Complicated Urinary Tract Infection; Pyelonephritis; Antimicrobial; Cephalosporin; Intravenous
MeSH Terms: conditions — Pyelonephritis | interventions — ceftolozane; Ceftazidime

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): CXA-101
  Interventions: Drug: CXA-101
- 2 (Active Comparator): Ceftazidime
  Interventions: Drug: Ceftazidime

INTERVENTIONS:
Drug: CXA-101 — intravenous
  Arms: 1
Drug: Ceftazidime — intravenous
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of intravenous CXA 101 and comparator in complicated urinary tract infection

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, prospective, randomized, double-blind, comparative efficacy and safety study of IV CXA 101 versus IV ceftazidime for 7 to 10 days.

Subjects are followed up 6 to 9 days after the last dose of study drug to assess clinical signs and symptoms of infection. A Late Follow Up evaluation (21 to 28 days after the last dose of study drug) occurs for those subjects who respond to therapy. The primary assessment of effectiveness is the microbiological response (the eradication at post-therapy of the infectious organism identified at the start of study). An additional assessment of efficacy includes the overall clinical response, which is described as cured, improved, or failed. Safety assessments include the incidence of adverse events throughout the study, clinical laboratory tests (hematology, serum chemistry, and urinalysis) and physical examinations at the start of the study and post-therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 to 90 years of age, inclusive.
2. Pyuria (white blood cell [WBC] count > 10/µL in unspun urine or ≥ 10 per high power field in spun urine)
3. Clinical signs and/or symptoms of cUTI, either of:

   a. Pyelonephritis, as indicated by both of the following: i. Fever (oral temperature ≥ 37.8°C); ii. Flank pain or costovertebral angle tenderness;

OR

b. Complicated lower UTI, as indicated by both of the following: i. At least one of the following new or worsening symptoms:

* Dysuria;
* Frequency;
* Suprapubic pain;
* Urgency

ii. At least one of the following complicating factors:

* Male gender;
* Current bladder instrumentation or indwelling urinary catheter that is expected to be removed during the course of IV study drug administration;
* Obstructive uropathy that is expected to be medically or surgically treated during the course of IV study drug administration;
* Urogenital surgery within 7 days preceding administration of the first dose of study drug;
* Functional or anatomical abnormality of the urogenital tract including anatomic malformations or neurogenic bladder with voiding disturbance of at least 100 mL residual urine.

Exclusion Criteria

1. Documented history of any hypersensitivity or allergic reaction to any β-lactam antibacterial
2. Concomitant infection requiring systemic antibacterial therapy in addition to IV study drug therapy at the time of randomization. Drugs with only gram-positive activity (e.g. vancomycin, linezolid) are allowed
3. Complete, permanent obstruction of the urinary tract
4. Confirmed (at time of randomization) fungal urinary tract infection (with ≥ 103 fungal CFU/mL)
5. Suspected or confirmed perinephric or intrarenal abscess
6. Suspected or confirmed prostatitis
7. Known ileal loop or vesico-ureteral reflux
8. Women who are pregnant or nursing

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2009-06-30 (Actual); Primary Completion 2010-02-25 (Actual); Study Completion 2010-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Haidar, MD, Principal Investigator — Mississippi Medical Research, LLC; Ryszard Gellert, MD, Principal Investigator — Szpital Bielański im.Ks. Jerzego Popiełuszki Samodzielny Publiczny Zakład Opieki Zdrowotnej IV Kliniczny Oddzial Chorób Wewnętrznych i Pododdział Nefrologiczny; Florian Wagenlehner, MD, Principal Investigator — Uniklinikum Giessen
Locations (21):
- United States (7):
  - Healthcare Partners Medical Group, Los Angeles, California
  - Compass Research, LLC, Orlando, Florida
  - Atlanta Institute for Medical Research, Inc., Decatur, Georgia
  - Infectious Disease of Indiana, PSC, Indianapolis, Indiana
  - Mississippi Medical Research, LLC, Picayune, Mississippi
  - Great Falls Clinic, LLP, Butte, Montana
  - Remington-Davis, Inc. Clinical Research, Columbus, Ohio
- Germany (7):
  - Kreiskrankenhaus Backnang, Backnang
  - URO Forschungs GmbH, Berlin
  - Uniklinikum Giessen, Giessen
  - Evangelisches Krankenhaus Giessen Urologie, Giessen
  - Universitätsklinikum Schleswig Holstein Campus Lübeck, Lübeck
  - Brüderkrankenhaus St. Josef Paderborn, Paderborn
  - Urologische Klinik Dr. Castringius München-Planegg, Planegg
- Poland (7):
  - Samodzielny Publiczny Szpital Kliniczny nr 4 Katedra i Klinika Nefrologii, Lublin
  - Wojewódźki Szpital Specjalistyczny nr 1 Oddział Chorób Wewnętrznych, Tychy
  - Szpital Bielański im.Ks. Jerzego Popiełuszki Samodzielny Publiczny Zakład Opieki Zdrowotnej IV Kliniczny Oddzial Chorób Wewnętrznych, Warsaw
  - Szpital Kliniczny Dzieciątka Jezus-Centrum Leczenia Obrażeń Klinika Urologii Ogólnej, Onkologicznej Czynnościowej, Warsaw
  - Szpital Praski p.w. Przemienienia Pańskiego Samodzielny Publiczny Zakład Opieki Zdrowotnej ll Oddział Wewnętrznych, Warsaw
  - Wojewódźki Szpital Specjalistyczny Oddział Nefrologiczny, Wroclaw
  - Samodzielny Publiczny Szpital Wojewódźki im. Papieża Jana Pawła ll Oddział Wewnętrznych Nefrologiczno-Endokrynologiczny ze Stacją Dializ, Zamość

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two subjects, one in each arm, did not receive treatment.
Groups:
- CXA-101: CXA-101: intravenous 1000 mg every 8 hours
- Ceftazidime: Ceftazidime: intravenous 1000 mg every 8 hours
Period: Overall Study
Arm/Group | CXA-101 | Ceftazidime
Started | 85 | 42
Completed | 81 | 39
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Received concomittant therapy | 2 | 0
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CXA-101 | Ceftazidime | Total
Number analyzed (Participants) | 85 | 42 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (19.78) | 62.7 (19.74) | 58.8 (19.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 16 | 58
  Male | 43 | 26 | 69

OUTCOME MEASURES:

1. Primary Outcome: Microbiological Response at the Test of Cure (TOC) Visit in the Microbiological Modified Intent-to-Treat (mMITT) Population
Description: Microbiological response is eradication for each baseline pathogen
Time Frame: TOC; 6-9 days after last study drug administration
Population: mMITT: Treated patients, with baseline pathogen.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CXA-101 | Ceftazidime
Number analyzed (Participants) | 65 | 38
percentage of patients | 83.1 [71.7 to 91.2] | 76.3 [59.8 to 88.6]
Statistical Analysis 1: Comparison: CXA-101 vs Ceftazidime; Test type: Superiority or Other; Risk Difference (RD) = 6.8

2. Primary Outcome: Microbiological Response at the TOC Visit in the Microbiologically Evaluable (ME) Population.
Description: Microbiological response is eradication for each baseline pathogen
Time Frame: TOC; 6-9 days after last study drug administration
Population: ME: Treated patients, with baseline pathogen, complied with protocol.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CXA-101 | Ceftazidime
Number analyzed (Participants) | 55 | 27
percentage of patients | 85.5 [73.3 to 93.5] | 92.6 [75.7 to 99.1]
Statistical Analysis 1: Comparison: CXA-101 vs Ceftazidime; Test type: Superiority or Other; Risk Difference (RD) = -7.1

ADVERSE EVENTS:
Arm/Group | CXA-101 | Ceftazidime
Serious Adverse Events (participants affected / at risk) | 1/85 | 0/42
Other Adverse Events (participants affected / at risk) | 33/85 | 16/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CXA-101 (N=85) | Ceftazidime (N=42)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CXA-101 (N=85) | Ceftazidime (N=42)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Arteriosclerotic retinopathy (Eye disorders) | 0 | 1
Retinal degeneration (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 8 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Gingival pain (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Feeling abnormal (General disorders) | 0 | 1
Infusion site erythema (General disorders) | 2 | 0
Infusion site extravasation (General disorders) | 2 | 0
Infustion site irritation (General disorders) | 3 | 0
Infusion site reaction (General disorders) | 1 | 1
Infustion site swelling (General disorders) | 2 | 0
Pyrexia (General disorders) | 3 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 5 | 0
Agression (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 4 | 0
Sleep disorder (Psychiatric disorders) | 6 | 2
Haematuria (Renal and urinary disorders) | 0 | 1
Renal cyst (Renal and urinary disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 1
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 1 | 1
Phlebitis (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The data generated in this clinical study are the exclusive property of the Sponsor and are confidential. Authorship on any primary publication of the results from this study will be based on contributions to study design, enrollment, data analysis, and interpretation of results.